CLINICAL TRIAL: NCT05719415
Title: Assessment of Recovery of Functional Capillary Surface Area in Patients Undergoing a Balloon Pulmonary Angioplasty for Chronic Thromboembolic Pulmonary Hypertension
Brief Title: Functional Pulmonary Capillary Surface Area in BPA for CTEPH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Dr David Langleben, Professor of Medicine, Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 00-034 (3)
Record Dates: First submitted 2023-01-30; First posted 2023-02-09 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Hypertension, Pulmonary; Pulmonary Thromboembolisms
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pre and post BPA (Experimental)
  Interventions: Other: Measurement of pulmonary functional capillary surface area

INTERVENTIONS:
Other: Measurement of pulmonary functional capillary surface area — Measurement of transpulmonary metabolism of trace injected doses of benzoyl-Phe-Ala-Pro

SUMMARY:
Chronic thromboembolic pulmonary hypertension [CTEPH] is caused by pulmonary emboli that have enlarged in pulmonary arteries and have become organized into the vessel wall. Many patients with CTEPH are treated with balloon pulmonary angioplasty [BPA] which mechanically opens the narrow pulmonary arteries. It is unclear how much downstream functional pulmonary capillary surface area [FCSA] is recovered during BPA. The investigators plan to measure FCSAIn CTEPH patients, before and after a session of BPA.

DETAILED DESCRIPTION:
Chronic thromboembolic pulmonary hypertension [CTEPH] affects approximately 3% of patients with a prior pulmonary embolism. In CTEPH patients, the acute pulmonary emboli do not resolve but instead become organized in the pulmonary artery walls causing physical luminal obstruction and impeding forward blood flow. Pulmonary vascular resistance rises, and right heart failure can ultimately develop. Currently, there are 3 therapeutic options for treating CTEPH: 1) pulmonary thromboendarterectomy involving surgical removal of the clots; 2) balloon pulmonary angioplasty involving opening of the narrow areas using angioplasty balloons; 3) medical therapy for distal disease using the soluble guanylate cyclase stimulator riociguat.

Balloon pulmonary angioplasty (BPA), depending on the number of narrow pulmonary artery segments that are opened, can provide immediate hemodynamic benefit in appropriate patients. Although the hemodynamics usually do not completely normalize after a single BPA session, cardiac output may increase and mean pulmonary artery pressure may fall. It is unclear how much pulmonary microvasculature must be restored to obtain this benefit, both in terms of number of segments, and in terms of the amount of downstream pulmonary microvasculature that must be regained.

The investigators have developed a technique in humans that assesses functional capillary surface area (FCSA). It involves measuring the metabolism of injected trace quantities of 3H-benzoyl Phe-Ala-Pro (BPAP), as the peptide passes through the lung circulation, and interacts with the capillary endothelial surface area. The investigators have established the range of normal in humans, studied the effects of exercise, and explored the reduction in FCSA in disease, including various types of pulmonary hypertension. Most germane to the present study, our previous work (Orfanos et al J Throm Hemostas 2008) demonstrated that the downstream capillary bed in CTEPH is functionally normal but FCSA is reduced because of upstream arteriolar blockage by organized thrombi. The average FCSA in untreated CTEPH is decreased by approximately 50%. Some of this FCSA should be immediately available to accept blood flow (recruitment) once the corresponding upstream segmental pulmonary artery is reopened by BPA.

Hypotheses:

1. The measured FCSA will immediately increase in CTEPH patients after BPA.
2. The amount of FCSA regained (recruited) will be proportional to the number of pulmonary arterial segments dilated.
3. The decrease in mean pulmonary arterial pressure towards normal may be a better indicator of FCSA regained than will be reduction in pulmonary vascular resistance.

Techniques:

All our routine techniques for BPA remain unchanged. The patients have a systemic arterial line and a pulmonary artery thermodilution catheter inserted for hemodynamic measurements prior to BPA, and the measurements are repeated after BPA. The only added procedure is that there will be 2 injections of 3H-BPAP via the "proximal" port of the thermodilution catheter, at the time of hemodynamic measurements pre-BPA (PRE) and post-BPA (POST). Systemic arterial blood will be collected at each timepoint for analysis of BPAP metabolism.

Recruitment and Consent:

The protocol has already been approved by the JGH IRB. Patients with newly diagnosed CTEPH who are deemed to be candidates for BPA will be approached in our Pulmonary Hypertension/CTEPH clinic. The research procedures and purpose will be explained and they will be given a consent form to review, and their questions will be answered. Should they agree to participate, the consent form will be signed and they will be included in the study.

Sample size:

Because BPAP metabolism will be measured pre and post BPA in the same patient, they will act as their own controls. The investigators are planning a study of a continuous response variable from matched pairs of study subjects. Prior data indicate that the baseline standard deviation of FCSA in the CTEPH population is 784. If the true FCSA difference in the mean response of matched pairs is 505 (33% increase in FCSA), the investigators will need to study 27 subjects to be able to reject the null hypothesis that this response difference is zero with probability (power) 0.9. If the mean response is 765 (50% increase), the investigators will need to study 13 subjects. The Type I error probability associated with this test of this null hypothesis is 0.05. The investigators will assess the magnitude of response after 10 subjects are completed and, based on that, reduce the n where possible. But the investigators have planned to study at least 40 subjects if needed.

ELIGIBILITY:
Inclusion Criteria:

* All patients eligible for balloon pulmonary angioplasty for chronic thromboembolic pulmonary hypertension

Exclusion Criteria:

* Treatment with angiotensin-converting enzyme inhibitors or angiotensin receptor blockers,
* Presence of patent foramen ovale

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2028-01-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in pulmonary functional capillary surface area | 4 hours
  Measurement of transpulmonary metabolism of benzoyl-Phe-Ala-Pro

CONTACTS AND LOCATIONS:
Locations (1):
- David Langleben, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No